CLINICAL TRIAL: NCT05578781
Title: Music-based Treatments and Pain: Underlying Mechanisms
Brief Title: Music-based Treatments and Pain: Underlying Mechanisms and the Beneficial Effects of Music-Based Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mark Jensen, Professor, School of Medicine: Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00014335; 1R21AT011577-01A1 (NIH)
Record Dates: First submitted 2022-10-06; First posted 2022-10-13 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Chronic Low-back Pain
Keywords: chronic; back pain
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Back Pain | interventions — Music Therapy; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial (RCT)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Music Therapy (Experimental): The Music Therapy (MT) group will participate in 1 live session of music therapy with a board certified Music therapist while wearing an EEG cap. Afterwards, they will complete a brief questionnaire about the experience and pain. They will also complete a brief questionnaire 24 hours later about lasting effects and pain
  Interventions: Behavioral: Music Therapy
- Music Medicine (Experimental): The Music Medicine (MM) group will participate in 1 audio session of music while wearing an EEG cap. Afterwards, they will complete a brief questionnaire about the experience and pain. They will also complete a brief questionnaire 24 hours later about lasting effects and pain
  Interventions: Behavioral: Music Medicine
- Control condition (Experimental): the Control group will participate in 1 session of an audio of text being read to them while wearing an EEG cap. Afterwards, they will complete a brief questionnaire about the experience and pain. They will also complete a brief questionnaire 24 hours later about lasting effects and pain
  Interventions: Behavioral: Control group
- Control group without low back pain (Active Comparator): This group will participate in 1 session of an audio of the music therapy session while wearing an EEG cap. Afterwards, they will complete a brief questionnaire about the experience and pain. They will also complete a brief questionnaire 24 hours later about the lasting effects and pain
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Music Therapy — Music Therapy is a music session with a live therapist and has been shown to reduce pain and anxiety. If effective the music medicine in this RCT will be used help design a full R01 study
  Arms: Music Therapy
Behavioral: Music Medicine — Music Medicine is an audio recorded music therapy session that will be played for the participant. This will be the same music session that will be played live in the music therapy session.
  Arms: Music Medicine
Behavioral: Control group — Control group will listen to an audio recording of text being spoken by the board certified music therapist
  Arms: Control condition; Control group without low back pain

SUMMARY:
The purpose of this study is to understand the mechanisms that underlie the beneficial effects of music-based treatments in individuals with moderate to severe chronic low back pain

DETAILED DESCRIPTION:
A growing body of research indicates that music may be used effectively for improving a variety of symptoms, including pain. However, little is known about the mechanisms that underlie the beneficial effects of music-based treatments. The primary objective of this R21 exploratory study is to evaluate the feasibility of performing a full R01 study in a sample of individuals with moderate to severe chronic low back pain to address knowledge gaps regarding the mechanisms of music-based treatments. To address the primary aims of this study, the investigators will conduct a 3-arm pilot trial in which individuals with chronic low back pain will be randomly assigned to one of three conditions: (1) live music played by a board-certified music therapist (Music Therapy), (2) audio recorded music (Music Medicine), or (3) audio of a person reading written text (n = 20 subjects per condition). In addition, 20 individuals without chronic pain will be enrolled and assigned to the Music Medicine condition.

An EEG assessment measuring brain oscillation spectral power will be conducted before and during a session of each experimental condition. Measures of pain intensity will be administered before and after the sessions. Low back pain was selected because it is among the most common, costly, and disabling chronic pain problems; including a non-pain sample will also allow us to determine if having chronic pain or not influences the effects of music on the primary mechanism variables. Effect sizes will be computed to evaluate (1) the effects of the treatments on frontal midline theta power and (2) the mediation effects of changes in frontal midline theta power on the pre- to post-session effects of the music conditions, relative to the control condition. The investigators will also investigate the differences between the three music conditions, compare the effects of Music Medicine on the mechanism variables as a function of having or not having chronic pain, and explore the extent to which the experimental conditions have lingering effects on pain intensity and secondary outcomes (depression, pain interference, and sleep quality) during the 24 hours after the experimental sessions. The investigators will also perform interviews and qualitative data analyses to identify additional unanticipated effects of the experimental conditions that would be worth examining more closely in a full R01 study. The findings from this study will be used to determine if a full R01 study to evaluate the mechanisms of music-based treatments is warranted, and to inform the design of such as study. This program of research will provide important foundational knowledge regarding the mechanisms of music-based interventions. Transferred to clinical care, this knowledge could help in patient-treatment matching which would enhance the overall effectiveness for music-based treatments and other non-pharmacological treatments that may operate via their effects on brain states, as measured by EEG.

ELIGIBILITY:
Inclusion Criteria for Chronic Low Back Pain sample:

* ≥18 years old
* Meets criteria for Chronic Low Back Pain (CLBP)
* Moderate to severe pain intensity on average (i.e., average pain in the past week ≥4 on the 0-10 NRS)
* Able to read, speak, and understand English

Inclusion criterion for the non-pain sample:

* ≥18 years old
* Able to read, speak, and understand English

Exclusion Criteria:

* Cognitive impairment that could interfere with study participation defined as ≥1 error on the 6-Item
* Presence of a psychiatric condition (e.g. significant suicidal ideation, active psychotic symptoms that would interfere with study participation
* Having a significant hearing disability that interferes with the potential participant's ability to hear music
* Having a health condition associated,per both chart review and self-report, with central nervous system damage (e.g., epilepsy, traumatic head injury, multiple sclerosis, Parkinson's).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Frontal Midline Theta Power | During the session
  Frontal midline theta power will be assessed using EEG assessment measuring brain oscillation spectral power for 5-min before and during each 20-min session.

SECONDARY OUTCOMES:
Duration of benefits | Pre-Intervention, immediately after intervention, as well as 24 hours later
  Estimated time of pain relief during the24 hours after the session, estimated using a 0-10 Numerical Rating scale.
Pain intensity | Pre-intervention and immediately after intervention
  Will be assessed using 0-10 Numerical Rating Scales (NRS).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jensen, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data that were used for the analyses presented in any paper published will be made available starting when the paper has been published to researchers who request it as long as they sign a data sharing agreement.
Supporting Information: Study Protocol, ICF
Time Frame: In order to obtain data, investigators who request it will be asked to indicate the specific analyses planned for those data, agree to not conduct any additional analyses not specified, agree not to share the data with others, and to destroy the data within a year of receipt or after the findings are published, whichever comes first.
Access Criteria: The PI of the project (Mark Jensen) will review all data requests.